CLINICAL TRIAL: NCT05407116
Title: Prospective Evaluation of Gastrointestinal and Genitourinary Side Effects of Pelvic Radiotherapy: Association Between Patient-Reported Outcomes and Clinician-Reported Outcomes With A View To Improving Quality of Care
Brief Title: Prospective Evaluation of Gastrointestinal and Genitourinary Side Effects of Pelvic Radiotherapy
Acronym: PROs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Joanne Alfieri, Associate professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-8347
Record Dates: First submitted 2022-02-23; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Radiotherapy Side Effects
Keywords: PROs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients receiving standard or hypofractionated radiotherapy for curative intent to a pelvic malignancy with an intended total dose of 25-60 Gy.
  Interventions: Other: NCI PRO-CTCAE Questionnaire / EORTC QLQ-C30 Questionnaire

INTERVENTIONS:
Other: NCI PRO-CTCAE Questionnaire / EORTC QLQ-C30 Questionnaire — PROs data will be collected prospectively via electronic questionnaires (PRO-CTCAE™), which is a patient-reported outcomes measurement system created to assess symptomatic toxicity in patients of cancer clinical research. PRO-CTCAE items evaluate frequency, severity, interference, amount, presence/absence symptoms. Each symptomatic adverse effect is measured by 1-3 features. GI items included nausea, vomiting, flatulence, bloating of the abdomen, constipation, diarrhea, abdominal pain, and loss of control of bowel movements. Urinary symptoms include the urge to urinate suddenly, frequency, urine colour change, loss of urine control (leakage).
  Patients will also self-report health-related quality of life (QoL) in real-time, electronic PRO questionnaires (EORTC QLQ CX24, EN 24, C30) about QoL. Question 29 and 30 ask the patients to rate their overall health and QOL respectively during the past week on a scale between 1-7, where one is equivalent to "very poor" and seven is "excellent."

SUMMARY:
Most patients who have pelvic radiotherapy (RT) as a treatment for cancer experience some degree of acute gastrointestinal (GI) and genitourinary (GU) toxicities. If physicians can anticipate, identify, and correctly manage symptoms, they can significantly improve patients' quality of life (QoL). Our study plans to enroll patients receiving standard or hypo-fractionated curative pelvic RT for the first time at the MUHC Radiation Oncology clinic. Patients will complete, through a mobile application (Opal) and in real-time, electronic patient-reported outcomes (PROs) questionnaires about acute GI/GU toxicities and quality of life (QoL). The treating physician will fill in the traditional intra-treatment forms simultaneously. The project's overall goal is to provide intra-treatment assessment tools to collect clinical information more relevant to the patients, improve patients' QoL, and triage clinically significant toxicities more efficiently.

DETAILED DESCRIPTION:
BACKGROUND: The classic endpoints in cancer clinical trials typically include tumour control rate, overall survival, or disease-free survival; however, it is becoming essential to consider the impact of cancer treatments on patients' quality of life (QoL) (1,2). Cancer researchers have used different methods to assess the effectiveness of therapeutic interventions according to their influences on health-related QoL (3,4). As with other cancer treatments, while radiotherapy (RT) can benefit cancer patients, its side effects can negatively impact QoL (5). Patients undergoing pelvic radiotherapy frequently develop acute gastrointestinal (GI) and genitourinary (GU) toxicities during treatment (6,7). If aware, the multidisciplinary team can manage ongoing problems patients are experiencing. This includes medical management, nutritional support and advice, and referral to other specialties (8). To date, most studies on toxicities from pelvic RT have used clinician-reported outcomes (CROs) for reporting intra-treatment assessments and guiding clinical practice and symptom management, but recent research shows that PROs better capture the quality of life issues that patients care about. In addition, consideration of patient-reported outcomes (PROs) leads to increased cancer treatment tolerance, reduced emergency room visits, earlier detection of recurrences, and improved survival (9,10). To our knowledge, there is no published prospective data assessing the association of CROs with PROs for GI/GU toxicities and QoL in patients undergoing radiation therapy to the pelvis. Therefore, there is a need to objectively examine how RT affects QoL in this patient group.

RATIONALE: Most patients who have radical pelvic RT as a treatment for cancer experience some degree of GI and GU toxicities (6,7). Anticipation, identification, and correct management of symptoms may significantly improve the QoL for those patients. This work aims to incorporate patient's voices during treatment and enhance the communication between patients and physicians, improve patients quality of life, and help early detection of adverse events All patients receiving standard or hypofractionated pelvic RT for the first time at the McGill University Health Centre Radiation Oncology clinic are eligible. Patients will complete, through a mobile application (Opal) and in real-time, validated electronic PRO questionnaires about acute GI/GU toxicities and QoL. These questionnaires will be administered at baseline, after each visit during RT, and at two subsequent time points, i.e., at two weeks and three-month follow-up visits. We will document data on any need for further assessment, prescriptions, emergency room visits, or admissions. The treating physician will fill in the traditional intra-treatment forms simultaneously.

ANALYSIS PLAN: Patient and treatment demographics will be summarized using proportions of categorical variables. We will perform a descriptive analysis for all GI/GU symptoms reported through patient and clinician questionnaires and assess the association between PROs and CROs over time using Somers' D statistic, Bowker's Symmetry test, and multilevel random effects regression models.

HYPOTHESIS: We hypothesize significant discordance between PROs and CROs when assessing GI/GU toxicities of pelvic RT and that CROs alone are insufficient in measuring GI toxicities as they fail to capture the impact on patients' quality of life. The study findings will assess the need for improved GI/GU symptom assessment and support the creation of a new algorithm that includes both patient and clinician input. In addition, physicians can influence the patients' quality of life by anticipating the problems and toxicities that need additional care, which they can appropriately expedite.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years or older
* Patients receiving standard or hypo-fractionated RT for curative intent to a pelvic malignancy
* Patients' ECOG performance status must be 0-2
* Patients should be able to give informed consent, read and understand English or French
* Patients should have access to the internet

Exclusion Criteria:

* Patients who have received prior pelvic radiation
* Patients who are at the end-of-life (expected survival less than six months)
* patients with significant cognitive dysfunction are excluded.
* patients included in other QoL studies, which may increase the patient burden and bias the answering of questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of collecting PROs and CROs for GI and GU toxicities prospectively and in real-time in a busy tertiary care cancer centre. | 18 weeks
  The attrition rate is well-defined as the number of patients who start reporting as a proportion of the number recruited, with causes of non-compliance. The questionnaire completion rate, which will be calculated as the number of questionnaires with at least five questions answered divided by the total number of potential questionnaires that could be administered through the study.
Assess the association between PRO and CROs over time | 18 weeks
  The primary outcome measures for assessing the association between PROs and CROs by comparing PRO-CTCAE symptom scores and clinician-reported CTCAE scores. Each PRO-CTCAE Symptom will be considered as a separate outcome, and correlated with its corresponding CTCAE Version 5.0 Term:

SECONDARY OUTCOMES:
Exploring the influence of baseline characteristics on treatment-related GI and GU symptoms | 18 weeks
  The influence of baseline characteristics such as age, gender, comorbidities (such as diabetes, hypertension, hyperlipidemia, pre-existing GI disease, pre-existing GU disease, and autoimmune disorders), current medications, smoking status and treatment-specific information such as prior chemotherapeutic agents, radiation dose and fractionation on treatment-related toxicity assessed using the PRO-CTCAE symptom scores.
Exploring the influence of baseline characteristics on health-related quality of life | 18 weeks
  The influence of baseline characteristics such as age, gender, comorbidities (such as diabetes, hypertension, hyperlipidemia, pre-existing GI disease, pre-existing GU disease, and autoimmune disorders), current medications, smoking status and treatment-specific information such as prior chemotherapeutic agents, radiation dose and fractionation on health-related quality of life will be assessed using the global quality of life score from the EORTC C30.
Assess whether PRO/CRO scores are associated with subsequent patient healthcare outcomes (changes in medications, ER visits, hospital admissions) | 18 weeks
  The ability to use PROs to triage patient symptoms by correlating PROs/CROs evolution of scores with management changes will be assessed by gathering data and clinical information such as changes in medications, ER visits, hospital admissions from patient files and correlating theses outcomes with the given scores

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laugsand EA, Sprangers MA, Bjordal K, Skorpen F, Kaasa S, Klepstad P. Health care providers underestimate symptom intensities of cancer patients: a multicenter European study. Health Qual Life Outcomes. 2010 Sep 21;8:104. doi: 10.1186/1477-7525-8-104. PMID 20858248
- [Background] Basch E, Jia X, Heller G, Barz A, Sit L, Fruscione M, Appawu M, Iasonos A, Atkinson T, Goldfarb S, Culkin A, Kris MG, Schrag D. Adverse symptom event reporting by patients vs clinicians: relationships with clinical outcomes. J Natl Cancer Inst. 2009 Dec 2;101(23):1624-32. doi: 10.1093/jnci/djp386. Epub 2009 Nov 17. PMID 19920223
- [Background] Budischewski K, Fischbeck S, Mose S. Quality of life of breast cancer patients in the course of adjuvant radiotherapy. Support Care Cancer. 2008 Mar;16(3):299-304. doi: 10.1007/s00520-007-0321-0. Epub 2007 Aug 7. PMID 17680279
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Yucel B, Akkas EA, Okur Y, Eren AA, Eren MF, Karapinar H, Babacan NA, Kilickap S. The impact of radiotherapy on quality of life for cancer patients: a longitudinal study. Support Care Cancer. 2014 Sep;22(9):2479-87. doi: 10.1007/s00520-014-2235-y. Epub 2014 Apr 12. PMID 24728584
- [Background] Chorbinska J, Krajewski W, Zdrojowy R. Urological complications after radiation therapy-nothing ventured, nothing gained: a Narrative Review. Transl Cancer Res. 2021 Feb;10(2):1096-1118. doi: 10.21037/tcr-20-2589. PMID 35116437
- [Background] Hafiz A, Abbasi AN, Ali N, Khan KA, Qureshi BM. Frequency and Severity of Acute Toxicity of Pelvic Radiotherapy for Gynecological Cancer. J Coll Physicians Surg Pak. 2015 Nov;25(11):802-6. PMID 26577965
- [Background] Denis F, Basch E, Septans AL, Bennouna J, Urban T, Dueck AC, Letellier C. Two-Year Survival Comparing Web-Based Symptom Monitoring vs Routine Surveillance Following Treatment for Lung Cancer. JAMA. 2019 Jan 22;321(3):306-307. doi: 10.1001/jama.2018.18085. PMID 30667494
- [Background] Lam E, Yee C, Wong G, Popovic M, Drost L, Pon K, Vesprini D, Lam H, Aljabri S, Soliman H, DeAngelis C, Chow E. A systematic review and meta-analysis of clinician-reported versus patient-reported outcomes of radiation dermatitis. Breast. 2020 Apr;50:125-134. doi: 10.1016/j.breast.2019.09.009. Epub 2019 Sep 19. PMID 31563429